CLINICAL TRIAL: NCT02720276
Title: Sms Guided Training After Acute Stroke: A Pilot Study
Brief Title: Sms Guided Training After Acute Stroke
Acronym: StrokeWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Birgit Vahlberg, Med Dr, RPT, Uppsala County Council, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UppsalaCC
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Acute Stroke
Keywords: stroke; exercise; walking; mobility
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training after acute stroke (Experimental): Intervention: Outdoor walking and strength training.
  Interventions: Other: Training after acute stroke

INTERVENTIONS:
Other: Training after acute stroke — Outdoor walking: Participants will receive daily training instructions via Short message Service (SMS) over 12 weeks. The walks are increased in frequency and intensity. The intensity are rated using the Borg scale to 12-15. The first 2 weeks begins with daily walks of 10 minutes. The last 4 weeks the walk training will partly be performed in intervals in combination with conventional outdoor walks. The interval training includes warming-up (5 minutes), fast walking for 4 minutes alternated with slower walking for three minutes. This is repeated 3 times, followed by cooling down for about five minutes. Strength training: to repeatedly get up from sitting. Number of repetitions will increase from 5-20 per set and will be performed daily in 3 sets with a short rest between each set.

SUMMARY:
The purpose of this exploratory study is to investigate how a predetermined outdoor walking program (12 weeks) is best delivered to individuals with stroke over 18 years, either by smartphone and the Short Message Service (SMS) or video link.

Furthermore, the aim is to investigate how the study design works in practice and determine the effects of the outdoor walking exercise program in combination with a leg exercise on physical functioning (walking capacity, gait speed, mobility and grip strength).

DETAILED DESCRIPTION:
Twenty community-living individuals in Uppsala municipality will be included and treated with a cross-over design. Ten individuals will initially receive exercise instructions to their smartphones via Short Message Service (SMS) for 6 weeks and after that instructions by a video link (6 weeks). Another 10 individuals will initially receive instructions by a video link and then switching to management with SMS after 6 weeks of training.

Intervention: Participants are supposed to perform an outdoor walking exercise program for 12 weeks. The walks should gradually increase in frequency and intensity, and is expected to start after discharge from the stroke department, after the assessment. The first 2 weeks start with daily walks. The walks will be conducted at a pace that increases the heart rate but still makes it possible to talk. The intensity and frequency of walks will progressively increase performed according to the Borg scale: 12-15, ie, moderate to strenuous. Participants will walk 5-7 days/week. Added to this is a strength exercise, which should be performed in connection with the walk training.

Methods: Questionnaires and medical records used for documentation of age, sex, comorbidity, blood pressure, medications and previous education.

Assessment of motor function, cognition, level of physical activity are only performed as screening at baseline measurements. Objective evaluation of the participants' adherence to the outdoor walking program will be measured with a training diary where the individual documents whether they have followed the training instructions.

Power analysis is not performed since this is an exploratory study. The investigators will analyze the data using an intention-to -treat. The investigators will also do a 'per-protocol analysis, where only participants who completed the training are included. Participants should have participated in at least 50% of the training sessions. All analyzes will be done using SPSS version 23 (IBM, Armonk).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. Verified ischemic cerebral infarction or intracerebral hemorrhage.
3. Sufficient walking capacity and motor function
4. Able to communicate in Swedish
5. Signed consent

Exclusion Criteria:

Are one or more of the following:

1. Subarachnoid bleeding
2. Insufficient cognition and impaired ability to understand instructions
3. Medical problems that make it unsuitable to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walk Test | change from baseline walking capacity to three months
  walking capacity

SECONDARY OUTCOMES:
Short Physical Performance Battery | change from baseline mobility to three months
  mobility
10 meters walk test | change from baseline gait speed to three months
  gait speed
Montreal Outcome Assessment | baseline
  cognitive function
Modified Rankin Scale | baseline
  motor function
Saltin Grimby Physical Activity Level Scale | baseline
  level of physical activity
Jamar hand dynamometer | change from baseline hand-grip strength to three months
  hand-grip strength
The Visual Analogue Rating Scale (VAS) | change from six baseline to three months.
  Report of how to deliver the best instructions.
The Visual Analogue Rating Scale (VAS) | change from baseline to three months.
  Report of how to deliver the best instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Vahlberg, Med Dr, RPT, Principal Investigator — VO Paramedicin

IPD SHARING:
Plan to Share IPD: No